CLINICAL TRIAL: NCT03960814
Title: Retrospective Cohort Study of All-Cause and Cardiovascular Mortality in Type 2 Diabetes Patients Using Basal Insulin Detemir and Glargine
Brief Title: A Study of All-Cause and Cardiovascular Mortality in Type 2 Diabetes Patients Using Basal Insulin Detemir and Glargine
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-4528; U1111-1233-0930 (Other: World Health Organization (WHO)); EUPAS29708 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: New users of basal insulins glargine and detemir
  Interventions: Drug: Insulin detemir

INTERVENTIONS:
Drug: Insulin detemir — No treatment will be given to the patients in relation to this study. Patients have been included in this study because they have been treated with insulin glargine or detemir prior to study initiation (2004 - 2018) and according to routine clinical practice at that time. The decision to initiate treatment with commercially available insulin detemir and glargine has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
This study will examine the influence of the basal insulins detemir and glargine on risk of cardiovascular death and death from all causes in patients treated by their general practitioner in United Kingdom (UK). The data for this study will be drawn from the Clinical Practice Research Datalink (CPRD) Register.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis (ever) of type 2 diabetes
* Prescription (ever) of basal insulins glargine or detemir
* Insulin-naïve until initiation of basal insulins glargine or detemir
* Aged 40 years or older at start of observation period

Exclusion Criteria:

* Diagnosis of type 1 diabetes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New users of basal insulins glargine and detemir
Sampling Method: Probability Sample
Enrollment: 12847 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Age at all cause death or censoring | Observation period 2004 - 2018
  Years
Age at death of cardiovascular disease | Observation period 2004 - 2018
  Years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bagsværd, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com